CLINICAL TRIAL: NCT03152318
Title: A Phase I Study of the Treatment of Recurrent Malignant Glioma With rQNestin34.5v.2, a Genetically Engineered HSV-1 Virus, and Immunomodulation With Cyclophosphamide
Brief Title: A Study of the Treatment of Recurrent Malignant Glioma With rQNestin34.5v.2
Acronym: rQNestin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Candel Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, E. Antonio Chiocca, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-557
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Malignant Glioma of Brain; Astrocytoma; Malignant Astrocytoma; Oligodendroglioma; Anaplastic Oligodendroglioma of Brain (Diagnosis); Mixed Oligo-Astrocytoma; Ependymoma; Ganglioglioma; Pylocytic/Pylomyxoid Astrocytoma; Brain Tumor; Glioma; Brain Cancer; Glioblastoma; Glioblastoma Multiforme
Keywords: Malignant Glioma; Brain Tumor; Glioblastoma; CAN-3110
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Disease; Ependymoma; Ganglioglioma; Brain Neoplasms; Glioma; Glioblastoma | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Phase I, open-label, single center, dose-escalation, triple-arm clinical trial of an oncolytic virus called rQNestin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A- rQNestin (Experimental): Arm A is rQNestin34.5v.2 treatment This study follows a standard 3+3 dose escalation design. Participants will not enroll to Arm B until the MTD or HTD has been met for Arm A.
  * Subjects with presumed radiologic evidence of recurrent malignant glioma will undergo stereotactic biopsy under monitored general or local anesthesia. Evidence of recurrent high grade or malignant must be found on frozen section for the person to receive administration of the agent.
  * rQNestin34.5v.2 Indicated dose as per cohort, Intratumor administration during surgery, single dose
  Interventions: Drug: rQNestin; Procedure: Stereotactic biopsy
- Arm B- rQNestin+CPA (Experimental): Arm B is rQNestin34.5v.2 treatment with Cyclophosphamide (CPA) pre-treatment This study follows a standard 3+3 dose escalation design. Participants will not enroll to Arm B until the MTD or HTD has been met for Arm A.
  * Cyclophosphamide one intravenous injection 2 days prior to procedure.
  * Subjects with presumed radiologic evidence of recurrent malignant glioma will undergo stereotactic biopsy under monitored general or local anesthesia. Evidence of recurrent high grade or malignant must be found on frozen section for the person to receive administration of the agent.
  * rQNestin34.5v.2 Indicated dose as per cohort, Intratumor administration during surgery, single dose
  Interventions: Drug: rQNestin; Drug: Cyclophosphamide; Procedure: Stereotactic biopsy
- Arm C- Multiple Dose rQNestin (Experimental): Arm C includes up to 6 intratumoral repeated doses of rQNestin34.5v.2, first in a cohort receiving 10^8 pfus per time point, followed by a cohort receiving 10^9 or 10^7 pfus per time point.
  * Arm C adds 2 cohorts of 12 subjects in an open-label clinical trial of rQNestin34.5v.2 administered at two dose levels
  * The injections are planned for days 0, 15, 30, 60, 90, and 120
  * Subjects with presumed radiologic evidence of recurrent malignant glioma will undergo stereotactic biopsy under monitored general or local anesthesia. Evidence of recurrent high grade or malignant must be found on frozen section for the person to receive administration of the agent.
  Interventions: Drug: rQNestin; Procedure: Stereotactic biopsy

INTERVENTIONS:
Drug: rQNestin — rQNestin is an oncolytic viral vector. It is administered via intratumoral injection during biopsy surgery.
  Other Names: rQNestin34.5v.2; CAN-3110
Drug: Cyclophosphamide — Cyclophosphamide is an immunomodulating agent. It is administered intravenously in a single dose 2 days (+/- 6 hrs) before surgery.
  Other Names: Cytoxan®; Neosar®
  Arms: Arm B- rQNestin+CPA
Procedure: Stereotactic biopsy — In both arms, subjects will undergo standard of care stereotactic biopsy in the intraoperative MRI operating room. The stereotactic needle will be placed stereotactically into the tumor bed using intraoperative MRI guidance to collect the biopsy, and again to administer the rQNestin oncolytic virus.

SUMMARY:
This research study is evaluating an investigational drug, an oncolytic virus called rQNestin34.5v.2. This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug as a possible treatment for this diagnosis of recurrent or progressive brain tumor.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug as a possible treatment for this diagnosis. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved rQNestin34.5v.2 as a treatment for any disease. This is the first time that rQnestin34.5v.2 will be given to humans.

The research drug, rQNestin34.5v.2, is an oncolytic viral vector made from the herpes simplex virus type 1 (HSV1). The large majority of humans already have regular HSV1 in their nervous system. Normally, this virus can cause cold sores in areas like the lips, fingers and genitals in humans by making copies of itself in normal healthy cells. In some cases, HSV1 can cause severe infection of the brain and liver and/or death. However, scientists have removed or changed parts of the rQNestin virus being used on this study so it can only make copies of itself in glioma cells and not normal healthy cells.

If it is effective, the rQNestin34.5v.2 drug will spread to a glioma cell, kill it, and then make a copy of itself and spread again. This should be repeated over and over until all glioma cells are reached. If rQNestin34.5v.2 moves into a normal brain cell, it should not grow and make copies, and therefore should not spread to other normal brain cells.

The purpose of this research study is to test if rQnestin34.5v.2 is safe to use in humans, and if it is effective in treating malignant glioma. This study is also looking for the highest dose of rQNestin34.5v.2 that can be given safely to people with malignant brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Frozen biopsy consistent with glioma by neuropathologist at the time of the first surgery in this longitudinal trial. Biopsy confirmation of glioma or infiltrative glioma at time of surgery will be acceptable, provided the subject has prior pathology confirmation of IDH wild-type glioma. Patients with reactive changes, gliosis or normal brain tissue only, without evidence of glioma at initial study surgery only will not receive study rQNestin34.5v.2 therapy and will be replaced. Confirmation of glioma at subsequent neurosurgical procedures beyond the initial surgery will not be required.
* Participants must have prior diagnosis of IDH wild-type glial tumor including GBM, grade 3 anaplastic astrocytoma or oligodendroglioma or or grade 2 astrocytoma with genetic features consistent with GBM, as confirmed by a neuropathologist or by a previous local pathology report. IDH wild-type designation may be based on negative immunohistochemistry (IDH1 R132H mutation) or next generation sequencing for patients with grade 4 tumor and by negative next-generation sequencing for those with grade 2 or 3 tumors. Patients with negative immunohistochemistry study for IDH1 R132H who are identified to have an alternative mutation of IDH1 or 2 are also not eligible.
* Prior history of external beam radiotherapy ≥ 5,000 cGy delivered to the tumor at least 4 weeks prior to OHRS registration. Participants over the age of 70 with prior history of hypofractionated external beam radiotherapy will also be accommodated, in accordance with NCCN guidelines.
* Prior history of temozolomide chemotherapy provided concurrent with external beam radiotherapy and after as per current standard of care. However, temozolomide is not required to have been provided concomitantly or after radiation if the patient had unmethylated MGMT promoter. At least 23 days must have passed from the last dose of temozolomide and first dose of rQNestin34.5v.2.
* For use of other investigational drug or other anti-tumor treatment, the following time periods must have elapsed from the projected start of scheduled study treatment: 4 weeks or 5 half-lives (whichever is shorter) from any investigational agent; 4 weeks from cytotoxic therapy (except 23 days for TMZ; 6 weeks from last dose for nitrosoureas); 12 weeks from completion of prior radiation therapy; 6 weeks from antibodies treatment; 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies; 1 day from NOVO-TTF (Optune®) or prior cancer vaccine therapy
* The initial recurrent or residual gadolinium-enhancing lesion to be treated must be at least 1.0 cm in diameter and less than or equal to 2 cm in greatest maximal diameter, as determined by MRI. The initially treated lesion must be located in non-eloquent cortex, defined as non-dominant temporal, frontal, or occipital lobe. If located in the dominant cortex, the lesion must be in the occipital lobe. For lesions in dominant or non-dominant lobes, there should be a judgment that the subject will be able to tolerate multiple injections and biopsies, based on sufficient distance from the enhancing edge and eloquent cortex defined as speech (dominant mid-to posterior temporal lobe, parietal lobe and frontal lobe: Broca's area), memory (hippocampus and mesial dominant temporal lobe), or sensorimotor cortex. Subsequent injections (injections at day 15, 30, 60, 90, 120) will not be subject to the limitations of the initially treated lesion detailed above.
* Normal hematological, renal and liver function as defined below before first injection: ANC ≥ 1000/mcL, platelets ≥100,000/mcL, PT or PTT <1.5 x institutional upper limit, Hemoglobin >9.0 g/dL, Total serum bilirubin ≤ 1.5 upper normal institutional limits, AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, and Serum creatinine ≤ 1.5 upper normal institutional limits OR Creatinine clearance ≥60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.
* Karnofsky Performance Score ≥70.
* Age ≥ 18 years;
* Ability to understand and the willingness to sign a written informed consent document;
* The effects of rQNestin34.5v.2 and cyclophosphamide on the developing human fetus are unknown. For this reason and because cytotoxic & immunomodulating agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation including 3 months following the study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation including 3 months following the study. Women of child-bearing potential must have a negative serum pregnancy test within 48 hours of study registration.
* No dexamethasone therapy for at least 14 days prior to the first rQNestin34.5v.2 inoculation. Patients who are on physiologic doses of corticosteroids for the treatment of adrenal insufficiency will be allowed to enroll.
* Ability to undergo MRI scanning with contrast;
* Have residual tumor or be at first or second relapse. Note: Relapse is defined as progression following initial therapy (i.e., radiation ± chemotherapy). For participants who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse. Residual tumor is defined as contrast-enhancing tumor that is present after the initial surgery, radiation, and chemotherapy.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (exceptions include but not limited to alopecia, laboratory values not listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).

Exclusion Criteria:

Participants who exhibit any of the following conditions prior to initiating study treatment will not be eligible for this study:

* Prior systemic malignancy requiring or expected to require more than surgical therapy within the past 24 months.
* Known chronic infections with HIV, hepatitis B or C; participants with a history of resolved Hepatitis A may be included in the trial.
* Participants with active viral, bacterial or fungal infection requiring concurrent antiviral or antibiotics.
* Subjects with active HSV-1 infection on current valacyclovir, acyclovir or ganciclovir therapy must be off treatment with any of these agents at least 7 days prior to surgery.
* Active, known, or suspected immunosuppressive disorders, such as acquired or congenital immune deficiency syndromes and autoimmune diseases.
* Unacceptable anesthesia risk
* Pregnant or lactating females who are breastfeeding.
* Participants who are receiving other investigational agents or immunotherapeutic agents during the period of rQNestin34.5v.2 longitudinal injections.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant active hepatic or renal disease, an active infection requiring systemic therapy, need for continuous systemic anticoagulation that cannot be stopped or psychiatric illness/social situations that would limit compliance with study requirements.
* Certain tumor sizes and locations are exclusionary: Participants with tumor ≤ 1 cm proximity to the ventricles will be allowed to enroll. However the study agent (rQNestin34.5v.2) may not be injected in any area that could lead to spillage into the ventricles regardless of where the tumor is located; Participants whose initial tumor size, location and rate of growth are deemed by the treating neurosurgeons and the CAC to not be able to tolerate the time period of expected longitudinal injections with biopsies, which could be as short as 15 days and as long as 120 days. This category would include tumors located in: a) dominant and non-dominant locations close to eloquent cortices (sensorimotor strip, speech and memory cortices), b) deep nuclear structures (caudate, putamen, thalamus), c) close proximity to corticospinal tracts (based on consensus of Clinical Advisory Committee); Participants with multifocal or multicentric tumors or tumors arising in the brain stem or spinal cord or diffuse leptomeningeal disease.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc.) within six months of registration.
* Has received anti-VEGF or anti-VEGFR targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc.)
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of registration.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of registration.
* Requires systemic anti-coagulation that cannot be halted for each intraoperative and peri-operative biopsy time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Minimum of 21 Days
  The primary objective is to determine the maximum tolerated dose of rQNestin34.5v.2 injected into recurrent malignant gliomas, with or without previous immunomodulation with cyclophosphamide.

SECONDARY OUTCOMES:
MRI Changes in Permeability | Evaluated every 2 months for 1 year
  Determine MRI alterations of permeability in injected sites using standard perfusion sequences.
MRI Changes in Volume | Evaluated every 2 months for 1 year
  Determine MRI alterations of cerebral blood volume in injected sites using standard sequences.
MRI Changes in Flow | Evaluated every 2 months for 1 year
  Determine MRI alterations of cerebral blood flow in injected sites using standard sequences.
Viral Shedding in Saliva | Evaluated up to day 56 for each subject
  Assess the shedding of rQNestin34.5v.2 in the saliva of subjects treated with rQNestin34.5v.2
HSV1 Viremia | Evaluated up to day 56 for each subject
  Assess the degree of HSV-1 viremia post rQNestin34.5v.2 administration
HSV1 Antibody Response | Evaluated up to day 56 for each subject
  Identify changes in HSV1 antibody response

CONTACTS AND LOCATIONS:
Overall Officials: E. Antonio Chiocca, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noh MH, Kang JM, Miller AA, Nguyen G, Huang M, Shim JS, Bueso-Perez AJ, Murphy SA, Rivera-Caraballo KA, Otani Y, Kim E, Yoo SH, Yan Y, Banasavadi-Siddegowda Y, Nakashima H, Chiocca EA, Kaur B, Zhao Z, Lee TJ, Yoo JY. Targeting IGF2 to reprogram the tumor microenvironment for enhanced viro-immunotherapy. Neuro Oncol. 2024 Sep 5;26(9):1602-1616. doi: 10.1093/neuonc/noae105. PMID 38853689
- [Derived] Ling AL, Solomon IH, Landivar AM, Nakashima H, Woods JK, Santos A, Masud N, Fell G, Mo X, Yilmaz AS, Grant J, Zhang A, Bernstock JD, Torio E, Ito H, Liu J, Shono N, Nowicki MO, Triggs D, Halloran P, Piranlioglu R, Soni H, Stopa B, Bi WL, Peruzzi P, Chen E, Malinowski SW, Prabhu MC, Zeng Y, Carlisle A, Rodig SJ, Wen PY, Lee EQ, Nayak L, Chukwueke U, Gonzalez Castro LN, Dumont SD, Batchelor T, Kittelberger K, Tikhonova E, Miheecheva N, Tabakov D, Shin N, Gorbacheva A, Shumskiy A, Frenkel F, Aguilar-Cordova E, Aguilar LK, Krisky D, Wechuck J, Manzanera A, Matheny C, Tak PP, Barone F, Kovarsky D, Tirosh I, Suva ML, Wucherpfennig KW, Ligon K, Reardon DA, Chiocca EA. Clinical trial links oncolytic immunoactivation to survival in glioblastoma. Nature. 2023 Nov;623(7985):157-166. doi: 10.1038/s41586-023-06623-2. Epub 2023 Oct 18. PMID 37853118
- [Derived] Otani Y, Yoo JY, Lewis CT, Chao S, Swanner J, Shimizu T, Kang JM, Murphy SA, Rivera-Caraballo K, Hong B, Glorioso JC, Nakashima H, Lawler SE, Banasavadi-Siddegowda Y, Heiss JD, Yan Y, Pei G, Caligiuri MA, Zhao Z, Chiocca EA, Yu J, Kaur B. NOTCH-Induced MDSC Recruitment after oHSV Virotherapy in CNS Cancer Models Modulates Antitumor Immunotherapy. Clin Cancer Res. 2022 Apr 1;28(7):1460-1473. doi: 10.1158/1078-0432.CCR-21-2347. PMID 35022322
- [Derived] Chiocca EA, Nakashima H, Kasai K, Fernandez SA, Oglesbee M. Preclinical Toxicology of rQNestin34.5v.2: An Oncolytic Herpes Virus with Transcriptional Regulation of the ICP34.5 Neurovirulence Gene. Mol Ther Methods Clin Dev. 2020 Mar 30;17:871-893. doi: 10.1016/j.omtm.2020.03.028. eCollection 2020 Jun 12. PMID 32373649